CLINICAL TRIAL: NCT05317598
Title: The Effect Of Posıtıve Psychotherapy-Based Courtesy And Honesty Psycoeducatıon On Effectıve Communıcatıon Skılls In Nursıng Students: The Key Model Of Courtesy And Integrıty
Brief Title: The Key Model Of Courtesy And Integrıty
Acronym: KMCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Kubra Gulırmak, Research assistant in psychiatric nursing department, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KÜBGÜ
Record Dates: First submitted 2022-03-10; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Psychotherapy; Communication
Keywords: Efective communication skills; positive psychotherapy; nursing students; psychoeducation; kindness and honesty.
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with a single-blind, pre-test post-test design.
Who Masked: Participant, Investigator
Masking Description: Participants in the pre-randomization study, two of the researchers, and the statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Students in the intervention group will be given a 5-week positive psychotherapy-based kindness and honesty psychoeducation.
  Interventions: Other: Kindness and honesty psychoeducation based on positive psychotherapy: The Key Model Of Courtesy And Integrity (KMCI)
- control group (No Intervention): Students in the control group will not receive any intervention during the 5-week period.

INTERVENTIONS:
Other: Kindness and honesty psychoeducation based on positive psychotherapy: The Key Model Of Courtesy And Integrity (KMCI) — It is an application that investigates the effect of kindness and honesty psychoeducation based on positive psychotherapy on effective communication skills of nursing students.
  Arms: Intervention group

SUMMARY:
Backround: Positive psychotherapy (PPT) divides conflicts into three. One of these conflicts is the key conflicts that occur frequently in daily life and arise from the unbalanced use of courtesy and honesty. Avoiding key conflicts depends on the balanced use of courtesy and honesty. Nursing students' balance of courtesy and honesty while communicating will reduce key conflicts and increase the level of effective communication skills. This is important in terms of making a significant contribution to the quality of nursing care. Objectives: This research was conducted to determine the effect of PPT-based kindness and honesty psychoeducation on the level of effective communication skills of nursing students. Design: The study is a randomized controlled, pretest-posttest design, and a single-blind study. Settings and participants: This research will conduct with 64 undergraduate nursing students who took a psychiatric nursing course. Methods: Students will divid into intervention and control groups by simple randomization method. "Personal information form and effective communication skills scale" will apply to the intervention and control groups. After the pre-measurements will apply, the intervention group received courtesy and honesty key (KMCI) psychoeducation for 5 weeks, and no intervention will apply to the control group. Afterwards, a post-test will apply to both groups.

Key words: Positive psychotherapy, effective communication skills, nursing students, psychoeducation, courtesy and honesty.

DETAILED DESCRIPTION:
Positive psychotherapy (PPT) is a humanistic-based, universal type of therapy derived from the positive psychology movement and developed by Nossrat Pessechkian in Germany in the 1960s. Although positive psychotherapy is basically based on analytical psychotherapies, it includes therapy approaches such as gestalt therapy and existential therapy and exhibits an eclectic approach with its unique methods. Among the basic concepts of positive psychotherapy are the capacities to love and to know, which are thought to be the two basic abilities that every person is born with. Later, he argues that these two basic abilities turn into other sub-skills over time and that many conflicts in daily life arise from the development of these abilities more or less. Conflicts have an important place in positive psychotherapy. It divides it into three main conflicts: real, fundamental and key conflict. The conflicts that the individual has experienced in daily life are real conflicts; Conflicts between primary or secondary abilities are expressed as basic conflicts. In this study, the conflict of courtesy and honesty, which is one of the key conflicts, is discussed. In terms of positive psychotherapy, the concept of honesty means that individuals are open. When individuals believe that openness and honesty are more important than being respectful of others, they openly express their opinions in a very open and direct way. This means that they use their honesty skills at a high level. Treating others with respect and courtesy is defined as courtesy. Courtesy is also a concept that is considered in the communication process. At this point, courtesy; It means to communicate by considering the feelings of the other people . Overuse of courtesy leads to the inability of the person to express himself honestly and to the role of victim, while overuse of the ability of honesty causes him to turn into a rudeness devoid of courtesy and to play an oppressive role. Therefore, the balanced use of courtesy and honesty skills is important. A courtesy that lacks honesty or a courtesy that does not contain honesty appears as a conflict in communication and interpersonal relations. Key conflicts between people are likely to occur frequently in daily life. Skills studies are carried out in positive psychotherapy in order to ensure the balanced use of honesty and courtesy skills in individuals. E.g; Raising awareness about the use of kindness and honesty skills and developing effective communication skills are the working subjects of positive psychotherapy.

Being able to communicate effectively is closely related to the balanced use of courtesy and honesty skills. Because, among the conditions of effective communication, it is emphasized that people should not play the role of oppressor or victim while expressing themselves. The ability to communicate effectively has a critical importance for professional groups such as nursing, which is based on human-to-human relations. It is very important for nurses to establish healthy and effective communication with the patient they care for, and to use their honesty and courtesy skills in a balanced way while establishing this communication. In the researches, it is seen that the skills of conflict management, problem solving and effective communication in the basic steps of effective communication are not at the desired level. It has been determined that they have difficulties in communicating especially with patients and their familie. However, in order to provide quality and qualified care to sick or healthy individuals with different needs; It is expected that they will be able to communicate effectively with them, use their courtesy-honest skills in a measured way, or gain the skills to manage crisis/conflict situations in a healthy way. In this context, students should have a high level of developing positive behaviors in interpersonal relations, establishing a balance of kindness and honesty in communication, overcoming conflicts easily, and thus establishing effective communication skills. For this reason, it is thought that the psychoeducation program will be effective in facilitating effective communication skills. When the literature is examined, it is seen that psychoeducation is very beneficial for students. When the international or national literature on positive psychotherapy is examined, it is seen that researches mostly consist of subjects such as creating life goals, depression, motivation to quit smoking, and creating a life purpose. However, it is seen that the studies on the key conflict issue are quite limited in the literature. It is also known that PPT has only just begun to enter the nursing literature. Therefore, this research is important both in terms of contributing to the nursing literature and in terms of its originality.

The aim of this study is to determine the effect of kindness and honesty key psychoeducation based on positive psychotherapy on effective communication skills in nursing students

ELIGIBILITY:
Inclusion Criteria:

* Being registered in the psychiatric nursing course and actively participating in the classes
* Being between the ages of 18-65
* Persons with computer/smartphone and internet access.

Exclusion Criteria:

* Students who did not meet the inclusion criteria,
* Did not complete the five-week pretest and posttest measurements,
* Did not actively continue the psychoeducation process,
* Did not have the necessary computer/smartphone and internet access to participate in the online psychoeducation program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
effective communication skills | 5 weeks
  According to the initial level of nursing students, the increase in the level of effective communication skills within the 5-week psychoeducation process was evaluated using the effective communication skills scale.

CONTACTS AND LOCATIONS:
Overall Officials: Eda ALBAYRAK, MSc, Study Chair — TC Erciyes University
Locations (1):
- Kübra Gülırmak, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rashid, T. (2015). Positive psychotherapy: A strength-based approach. The Journal of Positive Psychology, 10(1), 25-40.